CLINICAL TRIAL: NCT02031393
Title: Establishing First Trimester Sonographic, Biochemical and Clinical Markers for the Identification of High Risk Twin in the First Trimester
Brief Title: Establishing First Trimester Markers for the Identification of High Risk Twin
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: 217/13
Record Dates: First submitted 2014-01-08; First posted 2014-01-09 (Estimated); Last update posted 2014-01-31 (Estimated); Status verified 2013-12

CONDITIONS: Small for Gestational Age (Disorder); Pre-Eclampsia
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 9 Months
Biospecimen Retention: Samples Without DNA — Maternal serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- singelton pregnancy: will be followed 11-14 weeks and 19-28 weeks of gestation and after birth
- twin pregnancy: will be followed 11-14 weeks and 19-28 weeks of gestation and after birth

SUMMARY:
The purpose of this study is to determine whether we can establish different markers suc as mean arterial pressure , flow in the uterine arteries, biochemical markers in maternal blood and more un the first trimester, in order to screen for twin pregnancies that are more likely to develop adverse pregnancy outcome: early delivery, pre eclampsia or small fetuses.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women from 11 -14 weeks of gestation

Exclusion Criteria:

* nuchal thickness above 3 mm,
* Chronic hypertension,
* thrombophilia,
* Diabetes

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: pregnant women that will come to our first trimester clinic inorder to preform first trimester screeninig
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2009-09; Primary Completion 2014-01 (Actual); Study Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
The development of preeclampsia | after delivery
  the women will be approached after birth to asses whether they developed preeclampsia or pregnancy induced hypertension

SECONDARY OUTCOMES:
intra uterine growth restriction | after delivery

CONTACTS AND LOCATIONS:
Locations (1):
- Assaf Harofe obstetric department, Be’er Ya‘aqov, Zrifin, Israel